CLINICAL TRIAL: NCT05248568
Title: Effect of Core Training on Physical Fitness and Offensive Skills of Youth Male Basketball Players in China
Brief Title: Effect of Core Training on Physical Fitness and Offensive Skills, 12 Weeks Core Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Shengyao Luo, Principle Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: Luo Shengyao
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Experimental Myasthenia
Keywords: Core Training; Physical Fitness; Basketball Offensive Skills
MeSH Terms: conditions — Myasthenia Gravis, Autoimmune, Experimental

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Swiss ball (Experimental): Swiss ball practice can create an unstable environment and play an important role in promoting the development of muscle function and joint stability. It can effectively train the core muscles. Swiss ball practice will be involved in intermediate level training to develop participants' stability and muscle endurance。
  Interventions: Device: Core training
- Kettlebell (Experimental): Kettlebell training can strengthen the anti rotation ability of the trunk. For example, Kettlebell training has many actions like kettlebell swing. This movement is easy to cause imbalance in the human body, so they can further exercise the "trunk stability" and "anti rotation" ability required by athletes.
  Interventions: Device: Core training
- Barbell (Experimental): Barbell is a commonly used and multifunctional strength training instrument. It is usually used as the main instrument to develop the maximum muscle strength and muscle explosiveness. Therefore, this study will involve barbell practice in upper intermediate training and advanced level training
  Interventions: Device: Core training
- Medicine balls (Experimental): Medicine balls are often used to assist patients in injury recovery, rehabilitation and strength training, and play an important role in the field of sports medicine. Its special design and construction make training more functional and in line with the movement chain theory, such as throwing training, so the medicine ball is often used in explosive force and core training. Therefore, this study will involve medicine balls practice in upper intermediate training and advanced level training
  Interventions: Device: Core training

INTERVENTIONS:
Device: Core training — Core training lasts for 12 weeks, three times a week, one hour each time

SUMMARY:
The 12 week core training plan designed in this study is based on relevant literature and basketball characteristics. The training plan divides the training difficulty into four levels. The experimental group receives core training with different difficulties in 1-3 weeks, 4-6 weeks, 7-9 weeks and 10-12 weeks respectively.

DETAILED DESCRIPTION:
This paper designs the core training scheme based on the relevant literature and the characteristics of basketball. The training program of the experimental group lasts 12-weeks, 3 times per week, and 1 hour per training. The training program consists of four different difficulty levels, and the specific training contents are as follows: (1)Primary Level：Enhance trunk stability and prepare for more demanding core training (2)Intermediate Level：Continue to develop trunk stability and muscle endurance by increasing appropriate load (3)Upper-Intermediate Level：Increase the load weight, stimulate muscle hypertrophy and enhance the maximum strength level of muscle in the core area (4)Advanced-Level：Add more professional functional action modes in special sports, and develop the maximum strength and explosive force

The training contents as following:

1. Primary Level: In week 1-2 : Dead Bug (Body weight×15); Forearm Side Plank Crunch (Body weight×15); Plank Knee to Elbow (Body weight×15); Dynamic Bridge (Body weight×20); Single-Arm Dumbbell Bench press (10KG×15); All of these training with 2 sets and 60s recovery.

   Hanging Knee Hold (Body weight×60S); Elbow Plank (Body weight×90S); Side Plank (Body weight×60S); Supine planks (Body weight×90S); All of these training with 3 sets and 60s recovery.

   In week 3:

   Dead Bug (Body weight×15); Forearm Side Plank Crunch (Body weight×15); Plank Knee to Elbow (Body weight×15); Single-Leg Dynamic Glute Bridge (Body weight×20); Single-Arm Dumbbell Bench press (10KG×15); Hanging Knee Hold Body (weight×60S); Elbow Plank (Body weight×90S); Side Plank (Body weight×60S); Supine Planks (Body weight×90S); All of these training with 3 sets and 60s recovery.
2. Intermediate Level: In week 4: Barbell Hip Lift (65%1RM×15); Kneeling Cable Crunch (65%1RM×15); Stiff Leg Deadlifts (65%1RM×15); All of these training with 2 sets and 60s recovery.

   Swiss Ball Knee Tuck (Body weight×15); Kneeling Ab Wheel Rollouts(Body weight×15); Swiss Ball Bicycle Crunch (Body weight×15); All of these training with 3 sets and 60s recovery.

   Russian Twist (Body weight×25); Hanging Knee (Body weight×25); All of these training with 3 sets and 60s recovery.

   In week 5-6: Barbell Hip Lift (65%1RM×15); Kneeling Cable Crunch (65%1RM×15); Stiff Leg Deadlifts (65%1RM×15); Swiss Ball Knee Tuck (Body weight×20); Kneeling Ab Wheel Rollouts (Body weight×20); Swiss Ball Bicycle Crunch (Body weight×20); Russian Twist (Body weight×25); Hanging Knee (Body weight×25); All of these training with 3 sets and 60s recovery.
3. Upper-Intermediate Level： In week 7: Barbell Hip Lift (75%1RM×10); Barbell Bench Press (75%1RM×10); Stiff Leg Deadlifts (75%1RM×10); Barbell Bent-Over Row (75%1RM×10); All of these training with 3 sets and 90s recovery.

   Diagonal Plate Chop (15KG×15); Standing Ab Wheel Rollouts (Body weight×10); Barbell Hyper Extensions (15KG×15); Dumbbell Hanging Knee Raise (10KG×15); All of these training with 3 sets and 60s recovery.

   In week 8-9: Barbell Hip Lift (80%1RM×8); Barbell Bench Press (80%1RM×8); Stiff Leg Deadlifts (80%1RM×8); Barbell Bent-Over Row (80%1RM×8); All of these training with 3 sets and 120s recovery.

   Diagonal Plate Chop (20KG×10); Standing Ab Wheel Rollouts (Body weight×10); Barbell Hyper Extensions (20KG×10); Dumbbell Hanging Knee Raise (25KG×10); All of these training with 3 sets and 60s recovery.
4. Advanced-Level：In week 10: Landmine Rotation (25KG×15); Dead Ball Slam (5KG×10); Kettlebell Swing (25KG×15); Standing Chest Pass Medicine Ball (3KG×10); All of these training with 3 sets and 120s recovery.

Barbell Hip Lift (85%1RM×6); Barbell Bench Press (85%1RM×6); Stiff Leg Deadlifts (85%1RM×6); Barbell Bent-Over Row (85%1RM×6); All of these training with 3 sets and 180s-300s recovery.

In week 11-12: Landmine Rotation (30KG×12); Dead Ball Slam (8KG×8); Kettlebell Swing (30KG×12); Standing Chest Pass Medicine Ball (4KG×8); All of these training with 3 sets and 120s recovery.

Barbell Hip Lift (90%1RM×4); Barbell Bench Press (90%1RM×4); Stiff Leg Deadlifts (90%1RM×4); Barbell Bent-Over Row (90%1RM×4); All of these training with 3 sets and 180s-300s recovery.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-24 years
* Healthy
* Participants have received basketball training

Exclusion Criteria:

* Athletes who are systematically training their core strength
* Athletes with sports injuries unable to participate in core training

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-07-02 (Estimated)

PRIMARY OUTCOMES:
The Star Excursion Balance Test | week 1
  Before the SEBT can be performed, four strips of athletic tape will need to be cut to a length of 6-8 feet each. Two pieces will be used to form a'+', with the other two being placed over top to form an'x'so that a star shape is formed. It is important that all lines are separated from each other by a 45°angle.The goal of the SEBT is to maintain single leg stance on one leg standing in the centre of the star while reaching as far as possible with the contralateral leg.
  When using the right foot as the reaching foot, and the left leg to balance, the athlete should complete the circuit in a clockwise fashion. When balancing on the right leg, the athlete should perform the circuit in an anti-clockwise fashion.After they have completed a full circuit with each foot, a total of three times per leg.
  The test administrator should have recorded the reach distance of each successful attempt, with a pencil, in order to calculate the athlete's SEBT score after the test.
The Star Excursion Balance Test | week 6
  Before the SEBT can be performed, four strips of athletic tape will need to be cut to a length of 6-8 feet each. Two pieces will be used to form a'+', with the other two being placed over top to form an'x'so that a star shape is formed. It is important that all lines are separated from each other by a 45°angle.The goal of the SEBT is to maintain single leg stance on one leg standing in the centre of the star while reaching as far as possible with the contralateral leg.
  When using the right foot as the reaching foot, and the left leg to balance, the athlete should complete the circuit in a clockwise fashion. When balancing on the right leg, the athlete should perform the circuit in an anti-clockwise fashion.After they have completed a full circuit with each foot, a total of three times per leg.
  The test administrator should have recorded the reach distance of each successful attempt, with a pencil, in order to calculate the athlete's SEBT score after the test.
The Star Excursion Balance Test | week 12
  Before the SEBT can be performed, four strips of athletic tape will need to be cut to a length of 6-8 feet each. Two pieces will be used to form a'+', with the other two being placed over top to form an'x'so that a star shape is formed. It is important that all lines are separated from each other by a 45°angle.The goal of the SEBT is to maintain single leg stance on one leg standing in the centre of the star while reaching as far as possible with the contralateral leg.
  When using the right foot as the reaching foot, and the left leg to balance, the athlete should complete the circuit in a clockwise fashion. When balancing on the right leg, the athlete should perform the circuit in an anti-clockwise fashion.After they have completed a full circuit with each foot, a total of three times per leg.
  The test administrator should have recorded the reach distance of each successful attempt, with a pencil, in order to calculate the athlete's SEBT score after the test.

CONTACTS AND LOCATIONS:
Overall Officials: Shengyao Luo, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Wuhan Sports University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Because this is my doctoral thesis and it has certain confidentiality, I won't share it until I finish my doctoral thesis.

REFERENCES:
- [Background] Willardson, J. M. (2013). Developing the core. Human Kinetics.
- [Background] Gordon AT, Ambegaonkar JP, Caswell SV. Relationships between core strength, hip external rotator muscle strength, and star excursion balance test performance in female lacrosse players. Int J Sports Phys Ther. 2013 Apr;8(2):97-104. PMID 23593547